CLINICAL TRIAL: NCT03443570
Title: A Multicenter Prospective Randomized Study of Rituximab Combined With Bortezomib Versus Rituximab in the Treatment of Newly Diagnosed Primary Immune Thrombocytopenia (ITP)
Brief Title: Rituximab Combining Bortezomib Versus Rituximab in Management of ITP
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shandong University (Other)
Collaborators: The Affiliated Hospital of Qingdao University (Other); Yantai Yuhuangding Hospital (Other)
Responsible Party: Principal Investigator, Ming Hou, Professor and Director, Shandong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTX and bortezomib in ITP
Record Dates: First submitted 2018-02-18; First posted 2018-02-23 (Actual); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Immune Thrombocytopenia; Purpura, Thrombocytopenic, Idiopathic
Keywords: immune thrombocytopenia; Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Thrombocytopenia | interventions — Rituximab; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- combination treatment group (Experimental): 100 enrolled patients are randomly picked up to take rituximab in combination with bortezomib at the indicated dose
  Interventions: Drug: Rituximab; Drug: Bortezomib
- control group (Active Comparator): 100 enrolled patients are randomly picked up to take rituximabalone at the indicated dose
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — given with a fixed dose of 500 mg administered as an intravenous infusion every two weeks, for 2 times totally
  Other Names: rituximab injection
Drug: Bortezomib — given subcutaneous injection at a fixed dose of 2.0 mg weekly, for 4 times totally
  Other Names: velcade
  Arms: combination treatment group

SUMMARY:
The project was undertaking by Qilu Hospital of Shandong University and other 2 well-known hospitals in China. In order to report the efficacy and safety of rituximab combining with bortezomib for the treatment of adults with immune thrombocytopenia (ITP), compared to rituximab alone .

DETAILED DESCRIPTION:
The investigators anticipate to undertaking a parallel group, multicentre, randomised controlled trial of 100 ITP adult patients from 3 medical centers in China. One part of the participants are randomly selected to receive rituximab (given with a fixed dose of 500 mg administered as an intravenous infusion every two weeks, for 2 times totally) combining with bortezomib (given subcutaneous injection at a fixed dose of 2.0 mg weekly, for 4 times totally), the others are selected to receive rituximab alone (given with a fixed dose of 500 mg administered as an intravenous infusion every two weeks, for 2 times totally). Platelet count, bleeding and other symptoms were evaluated before and after treatment, adverse events are also recorded throughout the study in order to report the efficacy and safety of the combination therapy compared to rituximab alone therapy for the treatment of adults with ITP.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the diagnostic criteria for immune thrombocytopenia.
2. Not previously used rituximab and bortezomid,untreated patients, may be male or female, between the ages of 18 ~ 80 years.
3. To show a platelet count < 30×10^9/L, and with bleeding manifestations.
4. Eastern Cooperative Oncology Group（ECOG）performance status ≤ 2.

Exclusion Criteria:

1. Received chemotherapy or anticoagulants or other drugs affecting the platelet counts within 3 months before the screening visit.
2. Current HIV infection or hepatitis B virus or hepatitis C virus infections.
3. Severe medical condition (lung, hepatic or renal disorder) other than ITP. Unstable or uncontrolled disease or condition related to or impacting cardiac function (e.g., unstable angina, congestive heart failure, uncontrolled hypertension or cardiac arrhythmia)
4. Female patients who are nursing or pregnant, who may be pregnant, or who contemplate pregnancy during the study period.
5. Have a known diagnosis of other autoimmune diseases, established in the medical history and laboratory findings with positive results for the determination of antinuclear antibodies, anti-cardiolipin antibodies, lupus anticoagulant or direct Coombs test.
6. Patients who are deemed unsuitable for the study by the investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-03-01 (Estimated); Primary Completion 2020-03-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of platelet response(continuous response rate) | up to 3 year per subject
  Complete Response:a sustained (≥ 3 months) platelet count ≥100×10^9/L;response: a sustained (≥ 3 months) platelet count ≥ 30×10^9/L without recurrence of thrombocytopenia;No response (NR): platelet count < 30 × 10^9/L or a less than two fold increase in platelet count from baseline or the presence of bleeding. Platelet count must be measured on two occasions more than a day apart.

SECONDARY OUTCOMES:
therapy associated adverse events | up to 3 year per subject
  The number and frequency of therapy associated adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Ming Hou, Dr, Principal Investigator — Shandong University
Locations (1):
- Qilu hospital, Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No